CLINICAL TRIAL: NCT05917561
Title: Efficacy and Tolerance of the Association of ANIFROLUMAB (300mg) IV Every Four Weeks and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo: a Randomized Double Blind Prospective, Non Comparative Proof of Concept Phase II Study
Brief Title: Efficacy and Tolerance of the Association of ANIFROLUMAB (300mg) IV Every Four Weeks and Phototherapy Versus Phototherapy in Adults With Progressive Vitiligo
Acronym: VITANI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2022/03
Record Dates: First submitted 2023-05-31; First posted 2023-06-26 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Vitiligo
Keywords: anifrolumab; vitiligo; phototherapy; randomized
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, non-comparative, phase II proof-of-concept trial involved patients with progressive vitiligo and uses one of the most common regimens in this phase of study. Assessment of the experimental treatment efficacy will be estimated only on the results obtained in the experimental treatment arm (Anifrolumab 300mg/month + narrowband UVB TL01 arm).
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) This is a double-blind study. To preserve the blinding of the study, a minimum number of sponsor personnel will see the randomization table and treatment assignments before the study is complete.
  All study assessments will be performed by study personnel who are blinded to the patient's treatment group.
  Except in clinical circumstances where unblinding is required, the patients, investigators, sponsor study team, and any personnel interacting directly with patients or investigative sites will remain blinded to Anifrolumab and placebo assignment until after completion of the Double-Blinded Treatment Period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy associated with active treatment (Experimental): Anifrolumab 300mg/infusion/month for 36 weeks + UVB TL01: 2 times a week during 24 weeks. (Phototherapy will be started 12 weeks after the beginning of anifrolumab)
  Interventions: Drug: Anifrolumab Infusion Product
- Phototherapy associated with placebo (Placebo Comparator): Placebo once a month infusion for 36 weeks + UVB TL01: 2 times a week during 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anifrolumab Infusion Product — Anifrolumab 300mg/month infusion for 36 weeks
  Arms: Phototherapy associated with active treatment
Drug: Placebo — Placebo once a month, infusion for 36 weeks
  Arms: Phototherapy associated with placebo

SUMMARY:
The purpose of this phase 2 study is to evaluate the effect and the safety of the combination of ANIFROLUMAB in combination with phototherapy in adult participants with non-segmental progressive vitiligo

DETAILED DESCRIPTION:
Treatment Strategy: Multicentric, parallel double blind randomized phase 2 prospective study comparing ANIFROLUMAB (300mg/month) + narrowband UVB TL01 versus placebo + narrowband UVB TL01 Follow-up of the study: patients included in this study will start ANIFROLUMAB 3 months before starting narrowband UVB TL01. Phototherapy will be performed twice a week during 6 months. Follow-up visit will be done at week 12, 24, 36 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Subject: male or female aged ≥ 18 years and ≤ 65 years
* Subject with body weight ≥ 40kg
* Diagnosis of non-segmental (symmetrical) vitiligo with a body surface area involved >5% excluding hands and feet
* Active non-segmental vitiligo is defined by:

Non-segmental vitiligo with new patches or extension of old lesions during the last 6 months AND Presence of hypochromic aspect under Wood's lamp examination and/or perifollicular hypopigmentation under Wood's lamp examination.

* Able to read, understand, and give documented (electronic or paper signature) informed consent
* Registered in the French Social Security
* Agree to discontinue the use of the following excluded medications/treatments for at least 4 weeks prior to randomization (Visit 2) and throughout the study: systemic steroids, phototherapy, methotrexate, cyclosporine, mycophenolate mofetil, and azathioprine.
* Agree to discontinue the use of the following excluded medications for at least 2 weeks prior to randomization (Visit 2) and throughout the study:

TCS or topical immune modulators (e.g., tacrolimus or pimecrolimus) Topical phosphodiesterase type 4 (PDE-4) inhibitor (e.g. crisaborole) Topical JAK inhibitor (e.g., tofacitinib or ruxolitinib) and/or any other investigational topical treatments.

* Patient characteristics
* Are male or nonpregnant, nonbreastfeeding female patients:

  1. Male patients must agree to use 2 forms of birth control (1 must be highly effective, see below) while engaging in sexual intercourse with female partners of childbearing potential while enrolled in the study and for at least 4 weeks following the last dose of investigational product.
  2. Female patients of childbearing potential must agree to use 2 forms of birth control, when engaging in sexual intercourse with a male partner while enrolled in the study and for at least 12 weeks following the last dose of investigational product.

     The following birth control methods are considered acceptable (the patient should choose 2 to be used with their male partner, and 1 must be highly effective):

     Highly effective birth control methods: oral, injectable, or implanted hormonal contraceptives (combined estrogen/progesterone or progesterone only, associated with inhibition of ovulation); intrauterine device (containing copper) or intrauterine system (e.g., progestin-releasing coil); or vasectomized male (with appropriate post vasectomy documentation of the absence of sperm in the ejaculate). Effective birth control methods: condom with a spermicidal foam, gel, film, cream, or suppository; occlusive cap (diaphragm or cervical/vault caps) with a spermicidal foam, gel, film, cream, or suppository; or oral hormonal contraceptives.
  3. Females of non-childbearing potential are not required to use birth control and they are defined as:

Women ≥60 years of age or women who are congenitally sterile, or Women ≥40 and <60 years of age who have had a cessation of menses for ≥12 months and a folliculostimulating hormone (FSH) test confirming non-childbearing potential (≥40 mIU/mL or ≥40 IU/L), or women who are surgically sterile (i.e., have had a hysterectomy or bilateral oophorectomy or tubal ligation).

* Patients fully vaccinated against COVID-19. A patient is considered fully vaccinated ≥2 weeks after receipt of the second dose in a 2-dose series (Pfizer-BioNTech and Moderna).
* Signed informed consent form (ICF)

Exclusion Criteria:

General exclusion criteria

* Segmental or mixed vitiligo
* Patients that are currently experiencing or have a history of other concomitant skin conditions (e.g., psoriasis or lupus erythematosus) that would interfere with evaluations of the effect of study medication on vitiligo
* Patients who are currently experiencing a skin infection that requires treatment, or who are currently being treated with topical or systemic antibiotics.
* Patients that have any serious concomitant illness that is anticipated to require the use of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring. (e.g., unstable chronic asthma).
* Patients with history of basal cell or squamous epithelial skin cancer or melanoma
* Presence of significant uncontrolled neuropsychiatric disorder, are clinically judged by the investigator to be at risk for suicide.
* Current alcohol, drug, or chemical abuse

Exclusion criteria related to concomitant medications

* Patients that have been treated with the following therapies:

  1. monoclonal antibody (e.g., ustekinumab, omalizumab, dupilumab) for less than 5 half-lives prior to randomization.
  2. received prior treatment with any oral JAK inhibitor (e.g., tofacitinib, ruxolitinib)
  3. received any systemic corticosteroid administered within 4 weeks prior to planned randomization or are anticipated to require systemic corticosteroids during the study.
  4. received any systemic treatment with Methotrexate, Azathioprine, Cyclosporine within 12 weeks prior to planned randomization
  5. have had an intra-articular corticosteroid injection within 4 weeks prior to planned randomization.
  6. have received more than 250 UV lights sessions
* Patients that are largely or wholly incapacitated permitting little or no self-care, such as being bedridden.

Exclusion criteria related to infection and malignancy risk factors

* Any underlying condition that predisposes the subject to infection, including history of/current human immunodeficiency virus (HIV) infection
* An HIV test must be performed. The result should be available within 30 days of randomisation, but prior to the second dose of investigational product administration (Visit 2/Week 4).

Confirmed positive test for hepatitis B serology for:

1. Hepatitis B surface antigen, OR
2. Hepatitis B core antibody (HBcAb) AND hepatitis B virus (HBV) DNA detected above the lower limit of quantitation Note: Patients who were HBcAb positive at screening were tested every 3 months for HBV DNA. To remain eligible for the study, the patient's HBV DNA levels must have remained below the limit of quantitation

   * Positive test for hepatitis C antibody
   * Any of the following:

     1. Clinically significant chronic infection (ie, osteomyelitis, bronchiectasis, etc) within 8 weeks prior to Inclusion Visit (chronic nail infections not causing open skin lesions are allowed)
     2. Any infection requiring hospitalisation or treatment with IV anti-infectives not completed at least 4 weeks prior to Inclusion visit
   * Any infection requiring IV or oral anti-infectives (including antivirals) within 2 weeks prior to Inclusion visit
   * Have evidence of active TB or latent TB:

     1. have evidence of active TB, defined in this study as the following: Documented by a positive PPD test (≥5 mm induration between approximately 48 and 72 hours after application, regardless of vaccination history), medical history, clinical features, and abnormal chest x-ray at screening. The QuantiFERON®-TB Gold test or TSPOT®.TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. Patients are excluded from the study if the test is not negative and there is clinical evidence of active TB.

        Exception: Patients with a history of active TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met. Such patients would not be required to undergo the protocol-specific TB testing for PPD, QuantiFERON®-TB Gold test, or T-SPOT® TB test but must have a chest x-ray at screening.
     2. have evidence of untreated/inadequately or inappropriately treated latent TB, defined in this study as the following: documented to have a positive PPD test (≥5 mm induration between approximately 48 and 72 hours after application, regardless of vaccination history), no clinical features consistent with active TB, and a chest x-ray with no evidence of active TB at screening; or PPD test is positive and the patient has no medical history or chest x-ray findings consistent with active TB, the patient may have a QuantiFERON®-TB Gold test or TSPOT® TB test (as available and if compliant with local TB guidelines). If the test results are not negative, the patient will be considered to have latent TB (for purposes of this study); or QuantiFERON®-TB Gold test or T-SPOT® TB test (as available and if compliant with local TB guidelines) may be used instead of the PPD test. If the test results are positive, the patient will be considered to have latent TB. If the test is not negative, the test may be repeated once within approximately 2 weeks of the initial value. If the repeat test results are again not negative, the patient will be considered to have latent TB (for purposes of this study). Exception: Patients who have evidence of latent TB may be enrolled if he or she completes at least 4 weeks of appropriate treatment prior to randomization and agrees to complete the remainder of treatment while in the trial.

Exception: Patients with a history of latent TB who have documented evidence of appropriate treatment, have no history of re-exposure since their treatment was completed, and have a screening chest x-ray with no evidence of active TB may be enrolled if other entry criteria are met.

Such patients would not be required to undergo the protocol specific TB testing for PPD, QuantiFERON®-TB Gold test, or TSPOT® TB test but must have a chest x-ray at screening.

* Safety exclusions labs
* At Screening (within 4 weeks before Week 0 [Day 1]), any of the following:

  1. Aspartate aminotransferase (AST) >2.0 × upper limit of normal (ULN).
  2. Alanine aminotransferase (ALT) >2.0 × ULN.
  3. Total bilirubin >1.5ULN (unless due to Gilbert's syndrome)
  4. Serum creatinine >2.0 mg/dL (or >181 μmol/L)
  5. Neutrophil count <1000/μL (or <1.0 × 109/L)
  6. Platelet count <25000/μL (or <25 × 109/L)
  7. Haemoglobin <8 g/dL (or <80 g/L),
  8. Glycosylated haemoglobin (HbA1c) >8% (or >0.08) at screening (diabetic subjects only) Note: Abnormal screening laboratory tests may be repeated ONCE on a separate sample before subject is declared a screen failure.
* Confirmed COVID-19: The Baseline Visit must be at least 14 days from onset of signs/symptoms or positive SARS-CoV-2 test; symptomatic subjects must have recovered, defined as resolution of fever without use of antipyretics and improvement in symptoms;
* Suspected COVID-19: Subjects with signs/symptoms suggestive of COVID-19, known exposure, or high risk behavior should undergo molecular (e.g., polymerase chain reaction [PCR]) testing to rule out SARS-CoV-2 infection or must be asymptomatic for 14 days from a potential exposure. Perioperative management of investigational product Surgery should be avoided during the study if clinically feasible, but is permitted. If a surgery becomes necessary during the study, it should be scheduled at least 4 weeks after the previous administration of investigational product.

For non-major surgery, the decision to withhold investigational product administration is at the Investigator's discretion.

For major surgery, investigational product administration can be resumed at the Investigator's discretion after all of the following criteria are met:

* External wound healing is complete, and
* Any postoperative antibiotic course is completed, and
* All acute surgical complications have resolved Blood donations Subjects should not donate whole blood, blood components or sperm until the completion of the follow-up period.

Other non-inclusion criteria

* Have hypersensitivity to anifrolumab or to any of the excipients.
* Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures.
* Are currently enrolled in any other clinical trial involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have participated within the last 30 days in a clinical study involving an investigational product. If the previous investigational product has a long half-life (2 weeks or longer), at least 3 months or 5 half-lives (whichever is longer) should be allowed between the end of the previous treatment and the inclusion.
* Have previously been randomized in this study or any other study investigating anifrolumab.
* Are investigator site personnel directly affiliated with this study and/or their immediate families. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Score with VASI score | Week 36
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.

SECONDARY OUTCOMES:
Score with VASI score | Week 12
  Change in percentage of repigmented Surface area 12 weeks after-inclusion, by using the VASI score at week 12.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study
Score with VASI score Extent Score (VES) | Week 24
  Change in percentage of repigmented Surface area 24 weeks after-inclusion, by using the VASI score at week 24.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Score with VASI score Extent Score (VES) | Week 48
  Change in percentage of repigmented Surface area 24 weeks after-inclusion, by using the VASI score at week 24.
  The VASI Score is used to assess the severity and extent of Vitilgo. VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study.
Face Vitiligo Aera Scoring Index (F-VASI) score | Week 12
  Mean variation in percentage of Face Vitiligo Area Scoring Index (F-VASI) score between baseline , week 12
Face Vitiligo Aera Scoring Index (F-VASI) score | Week 24
  Mean variation in percentage of Face Vitiligo Area Scoring Index (F-VASI) score between baseline , week 24
Face Vitiligo Aera Scoring Index (F-VASI) score | Week 36
  Mean variation in percentage of Face Vitiligo Area Scoring Index (F-VASI) score between baseline , week 36
Face Vitiligo Aera Scoring Index (F-VASI) score | Week 48
  Mean variation in percentage of Face Vitiligo Area Scoring Index (F-VASI) score between baseline , week 48
Number of Adverse Events (AE) and serious adverse events (SAE), as well as the proportion of discontinuation due to AEs and/or SAEs | Week 36
  AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related, that occurs after a subject provides informed consent. Abnormal laboratory values or test results occurring after informed consent constitute AEs only if they induce clinical signs or symptoms, are considered clinically meaningful, require therapy, or require changes in the study drug.
Evaluation of score Vitiligo European Task Force (VETF) | Week 12
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score Vitiligo European Task Force (VETF) | Week 24
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score Vitiligo European Task Force (VETF) | Week 36
  Variation of the score Vitiligo European Task Force (VETF) The VETF score is used to assess the severity and extent of vitiligo. The VETF assesses 3 dimensions of the disease in 5 areas (Head/neck, hands and feet, trunk, arms, legs) namely 1/ extent: percentage of vitiligo involvement estimated using the rule of nines, 2/ depigmentation severity grading (stage 0: normal pigmentation Stage 1: incomplete pigmentation , stage 2 complete depigmentation, stage 3: partial hair whitening <30% stage 4: complete hair whitening) and 3/ spreading (score O: similar limits, Score 1: progressive vitiligo; score -1: regressive vitiligo).
Evaluation of score of the Vitiligo Extent Score (VES) | Week 48
  Variation in percentage of the Vitiligo Extent Score (VES). The VES score is used to assess the severity and extent of vitiligo. Using the VES calculator www.vitiligo-calculator.com, investigator choose the pictures that best represent the patient's skin lesions and then the percentage of depigmented area is calculated.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 12
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 24
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 36
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Vitiligo Signs of Activity Score (VSAS) | Week 48
  Variation in percentage of the Vitiligo Signs of Activity Score (VSAS). The VSAS score is used to assess the activity of the disease. It is assessed by evaluating the number of location with at least one disease sign of activity.
Evaluation of score of the Dermatology Life Quality Index (DLQI) Global Impression of Change-Vitiligo (PhGIC-V) | Week 12
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) Global Impression of Change-Vitiligo (PhGIC-V) | Week 24
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) Global Impression of Change-Vitiligo (PhGIC-V) | Week 36
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of score of the Dermatology Life Quality Index (DLQI) Global Impression of Change-Vitiligo (PhGIC-V) | Week 48
  Variation of the score of the Dermatology Life Quality Index (DLQI). DLQI is a 10-item instrument, each item scored from 0 to 3 where higher scores correspond to worse symptom impact, full range from 0 to 30.
Evaluation of the score of the Skindex 29 | Week 12
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Week 24
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Skindex 29 | Week 36
  Variation of the score of the Skindex 29. SkinDex29 is a 30-item instrument, each item scored from 1 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 150.
Evaluation of the score of the Vitiligo Impact Patient Scale (VIP) | Week 48
  Variation of the score of the Vitiligo Impact Patient Scale (VIP). Vitiligo Impact Scale is a 12-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of the score of the Vitiligo Impact Patient Scale (VIP) | Week 12
  Variation of the score of the Vitiligo Impact Patient Scale (VIP). Vitiligo Impact Scale is a 12-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of the score of the Vitiligo Impact Patient Scale (VIP) | Week 24
  Variation of the score of the Vitiligo Impact Patient Scale (VIP). Vitiligo Impact Scale is a 12-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of the score of the Vitiligo Impact Patient Scale (VIP) | Week 36
  Variation of the score of the Vitiligo Impact Patient Scale (VIP). Vitiligo Impact Scale is a 12-item instrument, each item scored from 0 to 5 where higher scores correspond to worse symptom impact, full range from 0 to 145
Evaluation of the Vitiligo Noticeability Scale (VNS) | Week 12
  Variation of the VNS score. The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable. higher score corresponds to worse symptom impact
Evaluation of the Vitiligo Noticeability Scale (VNS) | Week 24
  Variation of the VNS score. The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable. higher score corresponds to worse symptom impact
Evaluation of the Vitiligo Noticeability Scale (VNS) | Week 36
  Variation of the VNS score. The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable. higher score corresponds to worse symptom impact
Evaluation of the Vitiligo Noticeability Scale (VNS) | Week 48
  Variation of the VNS score. The VNS is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. The participant was asked to respond to the following query: Compared with before treatment, how noticeable is the vitiligo now? Responses: (1) more noticeable, (2) as noticeable, (3) slightly less noticeable, (4) a lot less noticeable, and (5) no longer noticeable. higher score corresponds to worse symptom impact
Evolution of Physician's Global Impression of Change- Vitiligo (PhGIC-V) | Week 12
  Variation of the PhGIC-V. The PhGIC-V is a physician measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Physician's Global Impression of Change- Vitiligo (PhGIC-V) | Week 24
  Variation of the PhGIC-V. The PhGIC-V is a physician measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Physician's Global Impression of Change- Vitiligo (PhGIC-V) | Week 36
  Variation of the PhGIC-V. The PhGIC-V is a physician measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Physician's Global Impression of Change- Vitiligo (PhGIC-V) | Week 48
  Variation of the PhGIC-V. The PhGIC-V is a physician measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Patient's Global Impression of Change- Vitiligo (PaGIC-V) | Week 12
  Variation of the PaGIC-V. The PaGIC-V is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Patient's Global Impression of Change- Vitiligo (PaGIC-V) | Week 24
  Variation of the PaGIC-V. The PaGIC-V is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Patient's Global Impression of Change- Vitiligo (PaGIC-V) | Week 36
  Variation of the PaGIC-V. The PaGIC-V is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of Patient's Global Impression of Change- Vitiligo (PaGIC-V) | Week 48
  Variation of the PaGIC-V. The PaGIC-V is a patient-reported measure of vitiligo treatment success that is rated on a 5-point scale. Overall improvement: (1) much improved, (2)minimally improved, (3)no change), (4)minimally worse, (5)much worse. Higher score corresponds to worse symptom.
Evolution of the Total Physician Global Vitiligo Assessment (T-PhGVA) | Week 12
  Variation fo the T-PhGVA: The T-PhGVA is a physician measure of vitiligo treatment success that is rated on a 4-point scale: overall improvement: (0) no change, (1)limited extent, (2)moderate extent, (3)extensive, (4)very extensive). Higher score corresponds to worse evaluation
Evolution of the Total Physician Global Vitiligo Assessment (T-PhGVA) | Week 24
  Variation fo the T-PhGVA: The T-PhGVA is a physician measure of vitiligo treatment success that is rated on a 4-point scale: overall improvement: (0) no change, (1)limited extent, (2)moderate extent, (3)extensive, (4)very extensive). Higher score corresponds to worse evaluation
Evolution of the Total Physician Global Vitiligo Assessment (T-PhGVA) | Week 36
  Variation fo the T-PhGVA: The T-PhGVA is a physician measure of vitiligo treatment success that is rated on a 4-point scale: overall improvement: (0) no change, (1)limited extent, (2)moderate extent, (3)extensive, (4)very extensive). Higher score corresponds to worse evaluation
Evolution of the Total Physician Global Vitiligo Assessment (T-PhGVA) | Week 48
  Variation fo the T-PhGVA: The T-PhGVA is a physician measure of vitiligo treatment success that is rated on a 4-point scale: overall improvement: (0) no change, (1)limited extent, (2)moderate extent, (3)extensive, (4)very extensive). Higher score corresponds to worse evaluation
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | Day 1
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | Week 12
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.
Evaluation of blood inflammatory markers using immunofluorescence on skin biopsies and ELISA multiplex. | Week 36
  Expression of IFN-α, TNF-α, IFN-γ, IL-4, IL-5, IL-12, IL-13, IL-15, IL-17, IL-22, IL-23, IL-33 CXCL4, CXCL9, CXCL10, CXCL11, CXCL12, CXCL16, CCL20, soluble HSP70.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Bordeaux, Bordeaux
  - Centre Hospitalier Régional Le Mans, Le Mans
  - Centre Hospitalier Universitaire de Nice, Nice
  - Centre Hospitalier Universitaire de Toulouse, Toulouse

REFERENCES:
- [Background] Ezzedine K, Eleftheriadou V, Whitton M, van Geel N. Vitiligo. Lancet. 2015 Jul 4;386(9988):74-84. doi: 10.1016/S0140-6736(14)60763-7. Epub 2015 Jan 15. PMID 25596811
- [Background] Picardo M, Dell'Anna ML, Ezzedine K, Hamzavi I, Harris JE, Parsad D, Taieb A. Vitiligo. Nat Rev Dis Primers. 2015 Jun 4;1:15011. doi: 10.1038/nrdp.2015.11. PMID 27189851
- [Background] Whitton ME, Pinart M, Batchelor J, Leonardi-Bee J, Gonzalez U, Jiyad Z, Eleftheriadou V, Ezzedine K. Interventions for vitiligo. Cochrane Database Syst Rev. 2015 Feb 24;2015(2):CD003263. doi: 10.1002/14651858.CD003263.pub5. PMID 25710794
- [Background] Hamzavi I, Jain H, McLean D, Shapiro J, Zeng H, Lui H. Parametric modeling of narrowband UV-B phototherapy for vitiligo using a novel quantitative tool: the Vitiligo Area Scoring Index. Arch Dermatol. 2004 Jun;140(6):677-83. doi: 10.1001/archderm.140.6.677. PMID 15210457
- [Background] Boniface K, Seneschal J, Picardo M, Taieb A. Vitiligo: Focus on Clinical Aspects, Immunopathogenesis, and Therapy. Clin Rev Allergy Immunol. 2018 Feb;54(1):52-67. doi: 10.1007/s12016-017-8622-7. PMID 28685247
- [Background] Bertolotti A, Boniface K, Vergier B, Mossalayi D, Taieb A, Ezzedine K, Seneschal J. Type I interferon signature in the initiation of the immune response in vitiligo. Pigment Cell Melanoma Res. 2014 May;27(3):398-407. doi: 10.1111/pcmr.12219. Epub 2014 Feb 21. PMID 24438589
- [Background] Jacquemin C, Rambert J, Guillet S, Thiolat D, Boukhedouni N, Doutre MS, Darrigade AS, Ezzedine K, Blanco P, Taieb A, Boniface K, Seneschal J. Heat shock protein 70 potentiates interferon alpha production by plasmacytoid dendritic cells: relevance for cutaneous lupus and vitiligo pathogenesis. Br J Dermatol. 2017 Nov;177(5):1367-1375. doi: 10.1111/bjd.15550. Epub 2017 Oct 25. PMID 28380264
- [Background] Boukhedouni N, Martins C, Darrigade AS, Drullion C, Rambert J, Barrault C, Garnier J, Jacquemin C, Thiolat D, Lucchese F, Morel F, Ezzedine K, Taieb A, Bernard FX, Seneschal J, Boniface K. Type-1 cytokines regulate MMP-9 production and E-cadherin disruption to promote melanocyte loss in vitiligo. JCI Insight. 2020 Jun 4;5(11):e133772. doi: 10.1172/jci.insight.133772. PMID 32369451
- [Background] Boniface K, Jacquemin C, Darrigade AS, Dessarthe B, Martins C, Boukhedouni N, Vernisse C, Grasseau A, Thiolat D, Rambert J, Lucchese F, Bertolotti A, Ezzedine K, Taieb A, Seneschal J. Vitiligo Skin Is Imprinted with Resident Memory CD8 T Cells Expressing CXCR3. J Invest Dermatol. 2018 Feb;138(2):355-364. doi: 10.1016/j.jid.2017.08.038. Epub 2017 Sep 18. PMID 28927891
- [Background] Morand EF, Furie R, Tanaka Y, Bruce IN, Askanase AD, Richez C, Bae SC, Brohawn PZ, Pineda L, Berglind A, Tummala R; TULIP-2 Trial Investigators. Trial of Anifrolumab in Active Systemic Lupus Erythematosus. N Engl J Med. 2020 Jan 16;382(3):211-221. doi: 10.1056/NEJMoa1912196. Epub 2019 Dec 18. PMID 31851795
- [Background] Brown SR, Gregory WM, Twelves CJ, Buyse M, Collinson F, Parmar M, Seymour MT, Brown JM. Designing phase II trials in cancer: a systematic review and guidance. Br J Cancer. 2011 Jul 12;105(2):194-9. doi: 10.1038/bjc.2011.235. Epub 2011 Jun 28. PMID 21712822
- [Background] Ratain MJ, Humphrey RW, Gordon GB, Fyfe G, Adamson PC, Fleming TR, Stadler WM, Berry DA, Peck CC. Recommended changes to oncology clinical trial design: revolution or evolution? Eur J Cancer. 2008 Jan;44(1):8-11. doi: 10.1016/j.ejca.2007.09.011. Epub 2007 Nov 5. No abstract available. PMID 17981025